CLINICAL TRIAL: NCT03014700
Title: Repurposing of Fibrinogen Concentrate as a Cost-Effective and Safe Hemostatic Agent in Infants Undergoing Cardiac Surgery on Cardiopulmonary Bypass
Brief Title: Fibrinogen Concentrate vs Cryoprecipitate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Glyn David Williams, Professor, Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36374
Record Dates: First submitted 2016-12-02; First posted 2017-01-09 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2017-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryoprecipitate Arm (Active Comparator): Subject will be administered Cryoprecipitate to control bleeding after open heart surgery when randomized to Cryoprecipitate group
  Interventions: Biological: Cryoprecipitate
- Fibrinogen Concentrate Arm (Active Comparator): Subject will be administered Fibrinogen Concentrate to control bleeding after open heart surgery when randomized to Fibrinogen Concentrate group
  Interventions: Biological: Fibrinogen Concentrate

INTERVENTIONS:
Biological: Fibrinogen Concentrate — Subject will be administered Fibrinogen Concentrate to control bleeding after open heart surgery when randomized to Fibrinogen Concentrate group
  Arms: Fibrinogen Concentrate Arm
Biological: Cryoprecipitate — Subject will be administered Cryoprecipitate to control bleeding after open heart surgery when randomized to Cryoprecipitate group
  Arms: Cryoprecipitate Arm

SUMMARY:
One of the most common hemostatic derangements in pediatric open- heart surgery is an acute acquired hypofibrinogenemia. This compromises fibrin clot generation and platelet aggregation, resulting in increased bleeding and allogenic blood transfusions.

Currently, fresh frozen plasma and cryoprecipitate are used to supplement fibrinogen in pediatric cardiac patients. We propose that replacing cryoprecipitate with fibrinogen concentrate will be as effective in treating post-CPB bleeding and will decrease total blood product exposure when used as part of a blood transfusion algorithm.

We plan to include all patients undergoing cardiac surgery on CPB less than 12 months and a fibrinogen level <250mg/dL while on bypass.

We hope to demonstrate that fibrinogen concentrate is at least as effective as the standard of care in the management of peri- operative bleeding in neonatal patients undergoing cardiopulmonary bypass. If we are able to demonstrate that fibrinogen is at least as effective as the standard of care, then we would plan a multi-center trial to demonstrate the safety and efficacy of this medication. If we are able to demonstrate that fibrinogen concentrate is effective, fibrinogen concentrate could replace allogenic products and potentially decrease transfusion related morbidity in mortality in this population.

DETAILED DESCRIPTION:
Patients under 12 months of age requiring cardiopulmonary bypass surgery will be approached for the study. Patients with a pre- existing coagulopathy, including unexplained bleeding or history of clotting, will be excluded. Prior to the study beginning, patients will be randomized to our standard transfusion algorithm with cryoprecipitate or fibrinogen concentrate. As is standard of care, laboratory tests will be sent at standard times points

1. after the induction of anesthesia,
2. after initiation of bypass,
3. after separation from bypass and administration of protamine, and transfusion of either fibrinogen concentrate or cryoprecipitate
4. on arrival to the ICU. These laboratory tests include hematocrit, arterial blood gas, chemistry, thromboelastogram (TEG) and fibrinogen. Additional laboratory tests will be sent as indicated by the clinical scenario to determine transfusion requirements. For patients enrolled in the study, we will standardize the anesthetic management, cardiopulmonary bypass protocol, and transfusion thresholds in the operating room and ICU. We will collect demographic data, intraop and post-op laboratory values, bypass times, intraop and post op transfusion data, chest tube output, adverse events, and length of ventilation, ICU stay and hospital stay.

For patients randomized to the study arm (fibrinogen concentrate), the fibrinogen level measured on bypass will be used to calculate the appropriate dose of fibrinogen concentrate to achieve a level of 300mg/dL after separation from bypass. Fibrinogen concentrate will replace cryoprecipitate in our post-operative transfusion algorithm. If the patient has continued bleeding based on laboratory values and clinical situation, the patient will be given cryoprecipitate as a rescue measure. Patients not on the study protocol will receive our normal transfusion algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of at least 32 weeks of gestational age and infants up to 12 months of age with the diagnosis of congenital heart disease, requiring open heart surgery with cardiopulmonary bypass

Exclusion Criteria:

* Pre-existing coagulopathy, including unexplained bleeding or history of clotting

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glyn D Williams, MBChB, FFA, Principal Investigator — Stanford University; Laura Downey, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - Laura Downey, Emory, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Started | 30 | 30
Completed | 25 | 29
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 4 [2 to 5] | 4 [2 to 7] | 4 [2 to 7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 14 | 21 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 22 | 18 | 40
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Units of Intraoperative Allogenic Donor Transfusions (ADT) Administered During Procedure Through ICU Arrival.
Description: For our study, 1 donor exposure = 1 unit of blood product transfusion. A blood product includes red blood cells, fresh frozen plasma, cryoprecipitate, and platelets.
Time Frame: From administration of the drug during surgery to ICU arrival postoperatively (up to 24 hours)
Measure: Median (Inter-Quartile Range); unit: ADT units
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Number analyzed (Participants) | 30 | 30
ADT units | 5 [4 to 7] | 4 [3 to 5]

2. Secondary Outcome: Chest Tube Output
Description: Volume of chest tube drainage evaluated over first 24 hours post operatively
Time Frame: From administration end of surgery to 24 hours post operatively
Population: Participants who completed the protocol are included in the analysis
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Number analyzed (Participants) | 25 | 29
ml/kg | 18.05 [10.94 to 26.03] | 16.11 [12.56 to 25.00]

3. Secondary Outcome: Hours of Mechanical Ventilation
Time Frame: From administration of the drug during surgery to extubation in the ICU (up to 30 days)
Population: Participants who completed the protocol are included in the analysis
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Number analyzed (Participants) | 25 | 29
hours | 30.32 [18.68 to 98.73] | 27.10 [20.42 to 51.58]

4. Secondary Outcome: Length of Stay in Intensive Care Unit (ICU)
Time Frame: From administration of the drug during surgery to discharge from the ICU (up to 3 months)
Population: Participants who completed the protocol are included in the analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Number analyzed (Participants) | 25 | 29
days | 4.50 [2.00 to 6.00] | 3.00 [2.00 to 7.00]

5. Secondary Outcome: Length of Stay in Hospital
Time Frame: From administration of the drug during surgery to discharge from the hospital (up to 6 months)
Population: Participants who completed the protocol are included in the analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Number analyzed (Participants) | 25 | 29
days | 8.00 [5.00 to 19.00] | 7.00 [4.00 to 11.00]

6. Secondary Outcome: Count of Participants Who Died Within 30 Days Following Procedure
Time Frame: From administration of the drug to 30 days following surgery
Population: Participants who completed the protocol are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
Number analyzed (Participants) | 25 | 29
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Day of procedure through 30 days postoperatively or hospital discharge
Arm/Group | Cryoprecipitate Arm | Fibrinogen Concentrate Arm
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 4/30
Other Adverse Events (participants affected / at risk) | 8/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoprecipitate Arm (N=30) | Fibrinogen Concentrate Arm (N=30)
Chest Exploration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 — Unrelated to study treatment
Death (General disorders) | 0 | 1 — Unrelated to study treatment
Stroke (Nervous system disorders) | 1 | 0 — Unrelated to study treatment
Tamponade (Cardiac disorders) | 0 | 1 — Unrelated to study treatment
Thrombosis requiring Intervention (Vascular disorders) | 0 | 1 — Unrelated to study treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoprecipitate Arm (N=30) | Fibrinogen Concentrate Arm (N=30)
Infection (with positive culture within 14 days) (Infections and infestations) | 1 | 0 — Unrelated to study treatment
Repeat Surgery (less than 7 days) (Surgical and medical procedures) | 2 | 0 — Unrelated to study treatment
Arrhythmia requiring treatment (Cardiac disorders) | 6 | 5 — Unrelated to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03014700/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03014700/SAP_001.pdf